CLINICAL TRIAL: NCT03795909
Title: Ruxolitinib Combined With Dexamethasone for Pediatric Refractory and Secondary Hemophagocytic Lymphohistiocytosis
Brief Title: Ruxolitinib Combined With Dexamethasone for HLH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Research Institute of Pediatrics (Other Government)
Responsible Party: Principal Investigator, Yan Yue, Principal Investigator, Capital Research Institute of Pediatrics
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: HLH-DR
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Hemophagocytic Lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — ruxolitinib; Dexamethasone; Hormones

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib and Placebo (Experimental): Ruxolitinib 2.5 mg twice daily by oral
  Interventions: Drug: Ruxolitinib; Drug: Dexamethasone
- Placebo and Ruxolitinib (Placebo Comparator): Sugar pill 2.5 mg twice daily by oral
  Interventions: Drug: Ruxolitinib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib （2.5 mg twice daily for patients if the age<14 years and the weight <25kg，5 mg twice daily for patients if the age<14 years and the weight≥25kg, 10mg twice daily for patients if the age ≥14 years and<18 years）
  Other Names: Jakafi
Drug: Dexamethasone — Dexamethasone (10mg/m2.d) delayes for the first 2 weeks（form week 1 to 2),(5mg/m2.d) from week 3 to 4，(2.5mg/m2.d) from week 5 to 6），1.25mg/m2.d for week 7，and dropped off on week 8.
  Other Names: Hormone

SUMMARY:
A protocol named as "HLH-DR" for patients with refractory and secondary hemophagocytic lymphohistiocytosismay.

DETAILED DESCRIPTION:
A modified protocol about ruxolitinib combined with dexamethasone which includes oral ruxolitinib (2.5 mg twice daily for patients if the age<14 years and the weight <25kg，5 mg twice daily for patients if the age<14 years and the weight≥25kg, 10mg twice daily for patients if the age ≥14 years and<18 years）. Dexamethasone (10mg/m2.d) delayes for the first 2 weeks （form week 1 to 2），(5mg/m2.d) from week 3 to 4，(2.5mg/m2.d) from week 5 to 6），1.25mg/m2.d for week 7，and dropped off on week 8. Every 2 weeks, patients can be evaluated based the diagnosed index

ELIGIBILITY:
Inclusion Criteria:

* Secondary and refractory HLH.

Exclusion Criteria:

* Family HLH.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Severity of disease | 2 weeks
  Serum ferritin>2000ng/ml, disease actvie; serum ferritin<2000ng/ml, disease control;

SECONDARY OUTCOMES:
Axillary temperature | 2 weeks
  36<Axillary temperature<37.2, disease control; 37.2<Axillary temperature<38.2, disease partly control; Axillary temperature>38.2, disease active

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yue, MD, Principal Investigator — Capital Institute of Pediatrics, China
Locations (2):
- China (2):
  - Yan Yue, Beijing, Chaoyang District
  - Yan Yue, Beijing